CLINICAL TRIAL: NCT06043024
Title: Characteristics of Cytokine Response in Patients With Temporomandibular Disorders Treated With Occlusal Splint Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Renata Sikora, DMD, DMD, Assistant, Faculty of Dental Medicine and Health, Josip Juraj Strossmayer University of Osijek
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2158-61-46-23-90
Record Dates: First submitted 2023-09-08; First posted 2023-09-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Temporomandibular Joint Disorders
Keywords: prospective study; interventional study
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMD pain group (Experimental): The arm includes patients with TMP pain screening scores ≥ 3 and with diagnosis of myalgia, arthralgia, headache attributed to TMP and painful disc displacement (with and without reduction) according to Axis I diagnostic criteria for temporomandibular disorders (DK/TMP). Patients will be treated with a stabilizing occlusal splint made of hard acrylate resin, about 1.5 mm thick in the posterior teeth area with an incisal plateau for canine guidance.
  Interventions: Device: Stabilization occlusal splint

INTERVENTIONS:
Device: Stabilization occlusal splint — Patients will be treated with a stabilizing occlusal splint made of hard acrylate resin, about 1.5 mm thick in the posterior teeth area with an incisal plateau for canine guidance. OS will be made by the same dental technician in the dental laboratory.
  Other Names: occlusal appliance

SUMMARY:
The goal of this intervention study is to determine the effect of occlusal splint (OS) therapy on the concentration of inflammatory cytokines in serum and gingival crevicular fluid (GCF) in patients with temporomandibular disorders (TMDs).

Aims are:

* to determine cytokines level in GCF and serum before and after OS therapy
* to determine the degree of psychosocial dysfunction and oral health-related quality of life before and after OS therapy
* investigate the correlation between cytokines level in GCF and serum
* to determine the effect of OS on treatment outcomes, pain intensity, dysfunction, and psychosocial status of patients with painful TMD. Participants will be asked to complete self-assessment questionnaires, and GCF and blood samples will be collected before beginning of the OS therapy and at follow-up examinations one month and two months after.

DETAILED DESCRIPTION:
Temporomandibular disorder (TMD) is a multifactorial disease with complex etiopathogenesis. The main symptoms are persistent pain in the masticatory muscles and preauricular region, limitations in jaw function, and sounds in the temporomandibular joints. The most commonly used therapy is the occlusal splint (OS). The therapeutic effect of OS is attributed to various factors, however the exact mechanism is still unknown. One of the potential diagnostic methods is the use of molecular biomarkers. Studies have demonstrated a correlation between inflammatory cytokines and pain in TMD patients compared to healthy controls. Molecular biomarker levels can be determined from tissue samples and body fluids. Gingival crevicular fluid (GCF) is a serum exudate that enters the gingival sulcus from the gingival plexus of blood vessels and contains proteins, various cell types, electrolytes, cytokines, etc. Considering its composition, wide availability, non-invasive method, and speed of collection, GCF could be a new source of TMD biomarkers with potential diagnostic, prognostic, and therapeutic purposes.

Participants diagnosed with myalgia, arthralgia, headache attributed to TMP and/or painful disk displacement (with and without reduction) according to DC /TMD will be included in the study. Participants will be asked to complete self-assessment questionnaires: Graded Chronic Pain Scale (v2), Jaw Functional Limitation Scale-20, Patient Health Questionnaire-9, Genaral Anxiety Disorder-7, Patient Health Questionnaire-15, Oral Behaviors Checklist, Oral health Impact Profile, and Perceived Stress Scale-10. The occlusal splints will be fabricated from hard acrylic resin by the same dental technician in the dental laboratory. The GCF sample will be collected from the sulcus using sterile tweezers and sterile paper sticks and placed in an Eppendorf tube containing 250 µl of 0.9% NaCl solution. Blood samples will be collected in Vacutainers and stored at +4°C until centrifugation. For multicomplex quantitative analysis of proinflammatory cytokines (interleukin 1 beta (IL -1β), interleukin 6 (IL - 6), interleukin 7 (IL -7), interleukin 8 (IL -8), interleukin 13 (IL -13), tumor necrosis factor alpha (TNF-α)), adapted ProcartaPlex multiplex assays will be used.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* TMP pain screening scores ≥ 3
* patients with natural teeth
* diagnoses: myalgia, arthralgia, headache attributed to TMP and painful disc displacement (with and without reduction) according to axis I diagnostic criteria for temporomandibular disorders (DK/TMP)

Exclusion Criteria:

* degenerative joint disease and subluxation of the temporomandibular joint (TMJ)
* head trauma
* orofacial pain not associated with temporomandibular disorders
* patients with fixed or removable prostheses
* patients who are currently undergoing orthodontic therapy and/or using occlusal splints
* patients who used anti-inflammatory drugs and muscle relaxants 48 hours before data collection, and patients who use drugs with an impact on the immune system (such as antiproliferative immunosuppressants, corticosteroids and other immunosuppressants, antirheumatic drugs, DMARDs, anti-lymphocyte monoclonal antibodies and other immunomodulating drugs , antidepressants, antiepileptics)
* periodontitis
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Change in cytokines level (IL-1beta, IL-13, IL-6, IL-7, IL-8, TNF alpha) in circulating blood after stabilization occlusal splint therapy | Baseline, one month, three months
  Custom ProcartaPlex Multiplex assays will be used for multicomplex quantitative analysis of inflammatory mediators. The entire protocol will be carried out according to the instructions of the manufacturer of eBioscience, Affymetrix.
Change in cytokines level (IL-1beta, IL-13, IL-6, IL-7, IL-8, TNF alpha) in gingival crevicular fluid (GCF) after stabilization occlusal splint therapy | Baseline, one month, three months
  Custom ProcartaPlex Multiplex assays will be used for multicomplex quantitative analysis of inflammatory mediators. The entire protocol will be carried out according to the instructions of the manufacturer of eBioscience, Affymetrix.

SECONDARY OUTCOMES:
Change in pain free opening, maximum unassisted opening and maximum assisted opening after stabilization occlusal splint therapy | Baseline, one month, three months
  Measuring the distance using a ruler between the incisal edge of the reference mandibular and maxillary incisor. Patients will be asked to open their mouth without feeling pain, then to open as wide as possible even though it is painful and the examiner will try to stretch the mouth with fingers further if possible.
Change in pain intensity and pain-related disability after stabilization occlusal splint therapy | Baseline, one month, three months
  Pain intensity and pain-related disability will be calculated using version 2 of the Graded Chronic Pain Scale (GCPSv2) self-report questionnaire from Axis II of Diagnostic Criteria for Temporomandibular Disorders (DC/TMP) with 3 items for pain intensity, 4 items for function and one item for number of days of pain. Characteristic Pain Intensity (CPI) is calculated by taking the mean value of items 2-4 (current pain, worst pain, average pain) and then multiplying by 10. Interference score is a score derived from the computed mean of items 6-8 (daily activities, social activities, work activities) and multiplied by 10. The total Disability Points are calculated by the sum of Points for Disability Days and Points for Interference Score. Classification of Chronic Pain Grade: Grade 0-no TMD pain; Grade I- low-intensity pain, without disability; Grade II- high-intensity pain, without disability; Grade III- moderately limiting; Grade IV- severely limiting.
Change in oral health-related quality of life in TMD patients after stabilization occlusal splint therapy | Baseline, one month, three months
  Oral health-related quality of life will be measured using the oral health impact profile (OHIP-14) questionnaire. OHIP-14 is a 14-item questionnaire with answers rated on a 5-point Likert scale. The total score is the sum of all answered items and the scale ranges from 0 to 56. As the total score increases, the quality of life decreases.
Change in perceived stress levels in TMD patients after stabilization occlusal splint therapy | Baseline, one month, three months
  Perceived stress levels will be measured with the self-assessment questionnaire Perceived Stress Scale-10 (PSS). PSS is a 10-item instrument with answers rated on a 5-point scale. A total PSS score will be calculated as a sum of all items after four positively stated items (items 4, 5, 7, and 8) are reversed. Higher scores indicate higher levels of perceived stress.
Change in jaw function limitation in patients with TMD after stabilization occlusal splint therapy | Baseline, one month, three months
  Change in jaw function limitation will be determined using the self-assessment questionnaire Jaw Functional Limitation Scale-20 (JFLS-20) from Axis II of DC/TMD. JFLS-20 is a 20-item instrument. The total score can be calculated as a mean value of available items while subscale scores for each type of functional limitation are calculated: chewing: mean of items 1-6; mobility: mean value of items 7-10; verbal and non-verbal communication: mean value of particles 13-20.
Change in depressed mood in patients with TMD after stabilization occlusal splint therapy | Baseline, one month, three months
  Change in depressed mood will be determined using the self-assessment questionnaire Patient Health Questionnaire-9 (PHQ-9). The total score is obtained by the sum of all points. The scale ranges from 0-27 with cut-points at 5, 10, 15, and 20 representing mild, moderate, moderately severe, and severe depression, respectively.
Change in anxious feelings and behavior in patients with TMD after stabilization occlusal splint therapy | Baseline, one month, three months
  Change in anxious feelings and behavior will be determined using the self-assessment questionnaire Genaral Anxiety Disorder-7 (GAD-7). The total score is obtained by the sum of all points. The scale ranges from 0 to 21, with cut-points at 5, 10, and 15 representing mild, moderate, and severe anxiety, respectively.
Change in physical symptoms in patients with TMD after stabilization occlusal splint therapy | Baseline, one month, three months
  Change in non-specific physical symptoms will be determined using a 15-item self-assessment questionnaire Patient Health Questionnaire-15 (PHQ-15) from Axis II of DC/TMD. Individual answers are scored and their sum gives the final result. The scale ranges from 0 to 30, with cut-points at 5, 10, and 15 representing low, medium, and high physical symptoms, respectively.
Change in the presence of parafunctional behaviors in patients with TMD after stabilization occlusal splint therapy | Baseline, one month, three months
  Change in the presence of parafunctional behaviors will be determined using the self-assessment questionnaire Oral Behaviors Checklist (OBC) from Axis II of DC/TMD. Scoring can be calculated as the sum of questions with a non-zero response. The scale ranges from 0 to 62. A score of 0-16 represents normal behaviors; a score of 17-24 occurs twice as often in TMD patients than in healthy individuals; a score of 25-62 represents a risk factor for TMD.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Smolic, Professor, Study Director — Faculty of dental medicine and health Osijek, Josip Juraj Strossmayer University Osijek
Locations (1):
- Helath Center Osijek-Baranja county, Osijek, County of Osijek-Baranja, Croatia